CLINICAL TRIAL: NCT02719860
Title: A Chemoprevention Trial to Study the Effects of High Tea Consumption on Smoking Related Oxidative Stress
Brief Title: High Tea Consumption on Smoking Related Oxidative Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03-0014
Record Dates: First submitted 2016-03-08; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer Prevention
MeSH Terms: interventions — Tea

ARMS (3):
- Green tea (Experimental)
  Interventions: Dietary Supplement: Green tea
- Black tea (Experimental)
  Interventions: Dietary Supplement: Black tea
- Placebo tea (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo tea

INTERVENTIONS:
Dietary Supplement: Green tea — 4 cups/day of green tea for 6 months; each cup is prepared by brewing 2 tea bags in 12 oz of water
  Arms: Green tea
Dietary Supplement: Black tea — 4 cups/day of black tea for 6 months; each cup is prepared by brewing 2 tea bags in 12 oz of water
  Arms: Black tea
Dietary Supplement: Placebo tea — 4 cups/day of placebo tea for 6 months; each cup is prepared by brewing 2 tea bags in 12 oz of water
  Arms: Placebo tea

SUMMARY:
The overall objective of this study is to determine the effect of high tea consumption on biological markers of oxidative stress that mediate lung cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 85% and at least 25 pack-years of current or former smoking history.
* No diagnosis of internal cancer within the last 5 years or no chemotherapy or radiation for an internal cancer within the last 5 years.
* Meets the Southwest Oncology Group (SWOG) performance status criteria of 0-1.
* Not be pregnant or intending to get pregnant during the study period (women participants).
* Willing to drink 4 cups of tea (each cup will be brewed with 2 tea bags and 12 ounces of water) for 1-month run-in period and for the 6-month intervention period.
* Willing to refrain from consuming other tea or tea products starting one month before the placebo run-in period and for the entire study period (a total of 8 months)
* Willing to refrain from consuming more than one caffeinated product (coffee, soda..) starting one month before the placebo run-in period and for the entire study period (a total of 8 months).
* Subjects cannot take mega-doses of vitamins during the trial. This is defined as more than 400 IU of vitamin E, 200 ug of selenium, or 1 gm of vitamin C per day, or more than the tolerable upper limits of any other supplement as defined in the Dietary Reference Intake panels developed by the Food and Nutrition Board under the Institute of Medicine. Such vitamin therapy must be discontinued at least 2 weeks prior to study entry.

Exclusion Criteria:

* Subjects immunosuppressed by virtue of medication or disease.
* Serious concurrent illness that could interfere with study regimen.
* Subjects with a history of invasive cancer within the past 5 years.
* Subjects who are drinking more than 5 cups of non-herbal tea per week.
* Subjects who cannot or are unwilling to consume caffeinated beverages.
* Subjects unable to perform forced expiratory maneuver during spirometry testing.
* More than one acute emphysema exacerbation within the last 6 month -period .
* Subjects on oxygen.
* Women with positive urinary pregnancy test.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2003-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Post-intervention change in urinary 8-hydroxydeoxyguanosine | Baseline and 6 months
Post-intervention change in urinary 8-F2-isoprostanes | Baseline and 6 months